CLINICAL TRIAL: NCT00757198
Title: Requirement of Analgesics After Two Remifentanil Dosing Regimen in Cardiac Surgery.
Acronym: REMISYD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Pasi Lahtinen, PhD,MD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH5070206; EudraCT 2008-000597-21
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Pain
Keywords: pain, postoperative, opioid, PCA, cardiac surgery
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): remifentanil o.1 mcg/kg/min
  Interventions: Drug: remifentanil
- 2 (Active Comparator): remifentanil 0.3 mcg/kg/min
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — remifentanil infusion
  Arms: 1
Drug: remifentanil — remifentanil infusion
  Arms: 2

SUMMARY:
Prospective double blind study comparing two remifentanil dosing protocols (0.1 and 0.3 mcg/kg/min) during cardiac surgery. Main outcome measures are postoperative opioid requirements (PCA oxycodone) and postoperative pain (VAS, verbal rating scale).

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery bypass grafting patients

Exclusion Criteria:

* Psychiatric disorders, sleep apnea, cardiac insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid (oxycodone) consumption | Postoperatively 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pasi Lahtinen, MD, Study Director — Department of Anesthesiology and Intensive Care, Kuopio University hospital, Kuopio, Finland
Locations (1):
- Kuopio University hospital, Kuopio, Finland